CLINICAL TRIAL: NCT00350233
Title: MR Guided Focused Ultrasound Surgery of Metastatic Bone Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM002
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Bone Metastases
Keywords: Bone Tumors; Bone Cancer; Prostate Cancer; lung cancer
MeSH Terms: conditions — Bone Neoplasms; Prostatic Neoplasms; Lung Neoplasms

ARMS (1):
- ExAblate MRgFUS (Experimental)
  Interventions: Device: ExAblate 2000

INTERVENTIONS:
Device: ExAblate 2000

SUMMARY:
The objective of this trial is to evaluate the safety and effectiveness of MRgFUS in the treatment of metastatic bone tumors.

DETAILED DESCRIPTION:
Bone is the third most common organ involved by metastasic disease behind lung and liver. In breast cancer, bone is the second most common site of metastatic spread, and 90% of patients dying of breast cancer have bone metastasis. Breast and prostate cancer metastasize to bone most frequently, which reflects the high incidence of both these tumors, as well as their prolonged clinical courses.

Post cancer survival has increased with improvement in early detection and treatments. As a consequence, the number of patients developing metastatic bone disease during their lifetime has also increased. Patients with bone metastasis from breast cancer have an average 2-year survival from the time of presentation with their first bone lesion. In patients who die from breast, prostate, and lung cancer, autopsy studies have shown that up to 85% have evidence of bone metastases at the time of death.

Current treatments for patients with bone metastases are primarily palliative and include localized therapies (radiation and surgery), systemic therapies (chemotherapy, hormonal therapy, radiopharmaceutical, and bisphosphanates), and analgesics (opioids and non-steroidal anti-inflammatory drugs). Recently, radiofrequency ablation has been tested as a treatment option for bone metastases. The main goals of these treatments are improvement of quality of life and functional level. These goals can be further described: 1) Pain relief, 2) Preservation and restoration of function, 3) Local tumor control, 4) Skeletal stabilization.

The study hypothesis is that MRgFUS is a safe and potentially effective non-invasive treatment for metastatic bone tumors with a low incidence of co-morbidity. Based on the result of this study the Sponsor will initiate a larger study in an effort to approve metastatic bone tumors as an indication for its MRgFUS ExAblate device.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 and older
2. Patients who are able and willing to give consent and able to attend all study visits
3. Patients with histologically or cytologically confirmed malignant disease with a bone lesion that appears to be metastatic disease by clinical and or imaging techniques
4. Must have persistent pain from at least one site of bone metastases

   * Patient with VAS pain score ≥ 4, when VAS test taken without medication, OR
   * Patient taking pain-relieving medication for management of bone metastases.
5. Targeted tumor(s) are ExAblate device accessible
6. Targeted tumor(s) size is smaller than 8 cm in diameter
7. Patient whose lesion is on bone and is ≥ 10-mm from the skin.
8. Tumor(s) clearly visible by non-contrast MRI
9. Able to communicate sensations during the MRgFUS ExAblate treatment
10. At least 2 weeks since chemotherapy
11. At least 1 month since radiation therapy

Exclusion Criteria:

1. Diffuse skeletal tumoral spread as evaluated by imaging.
2. Patients who need pre-treatment surgical stabilization of the affected bony structure.
3. Targeted tumor is in weight bearing bones or impending fracture
4. Targeted tumor is in the vertebral column.
5. Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication
   * Patients with documented myocardial infarction within six months of protocol entry
   * Congestive heart failure requiring medication (other than diuretic)
   * Patients on anti-arrhythmic drugs
6. Severe hypertension (diastolic BP > 100 on medication)
7. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations (weight >250 pounds), etc.
8. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist)
9. ASA Score>2 (See "Definitions" below)
10. Extensive scarring in an area in the path of energy planned passage to the treatment area
11. Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
12. Patients on anti-coagulation therapy or those with an underlying bleeding disorder.
13. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 3 hrs.)
14. Patient whose lesion is < 10-mm from the skin
15. Patients with < 2-Weeks since chemotherapy
16. Patient with < 1-Month since radiation therapy
17. Patients with life expectancy < 6-Months
18. Patients with surgical stabilization of tumor site with metallic hardware

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Determine safety of MRgFUS of Bone Metastases | Within 1 month of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, M.D., Principal Investigator — University of California, San Diego; David Gianfelice, M.D., Principal Investigator — Toronto General Hospital
Locations (2):
- University of California at San Diego, La Jolla, California, United States
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- See also: Sponsor Web Page — http://www.insightec.com